CLINICAL TRIAL: NCT01165697
Title: Establishment of Biomarkers for Fabry Disease
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Deb Grzybowski, Research Assistant Professor, Ohio State University
Other Study IDs: 2009H0137
Record Dates: First submitted 2010-07-16; First posted 2010-07-20 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Fabry Disease
Keywords: Fabry Disease; vascular disease; storage endotheliopathy
MeSH Terms: conditions — Fabry Disease; Vascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fabry disease biomarker: Neuro-retinal fluorescein angiography (NRFA) exam will be administered once every 6 months for up to 3 years.
  Interventions: Other: Fluorescein angiography

INTERVENTIONS:
Other: Fluorescein angiography — Fluorescein angiography once every 6 months for 3 years

SUMMARY:
Fabry disease, an x-linked recessive lysosomal storage disease (LSD) is commonly recognized as a cause of renal failure in involved men and more recently recognized in women too. Women are involved in significant numbers and with complications, as are men, of vascular disease. This manifests as unexpected strokes in young adults. We have morphologic evidence that storage-endotheliopathy induced microvascular disease is the cause of cardiopathy and of cryptogenic strokes, and that storage endotheliopathy starts in early life, probably before birth. Based on our earlier work with other endotheliopathies such as diabetes mellitus, Susac syndrome, and hypertension, we will find and study patients using unique methods, neuro-retinal fluorescein angiography (NRFA), that we have developed for this purpose. These methods include NRFA to demonstrate capillary perfusion in the optic nerve head and retinal quadrants. We anticipate, based on our earlier experience with other endotheliopathies, that we will show more vascular pathology earlier than previously reported. Using epidemiologic and genetic tools we will find more patients than previously known or expected. It will offer opportunity for earlier diagnosis, prognosis, and response to enzyme replacement therapy.

We hypothesize that Fabry disease is a poorly recognized and poorly characterized cause of microvascular disease and cryptogenic strokes in young women and men. Neuroretinal capillary perfusion abnormalities in Fabry disease will be predictive of equivalent vascular disease in kidney, heart, brain and other organs, and further that it will be responsive to change induced by enzyme replacement therapy treatment.

DETAILED DESCRIPTION:
Specific Aims

Specific Aim 1. To demonstrate the specificity and sensitivity of the diagnostic capabilities of a neuroretinal examination which includes slit lamp and fundoscopy, and NRFA for the diagnosis of Fabry disease on a subject population of identified FD patients.

Specific Aim 2. To show capillary perfusion abnormalities in optic nerve and retina using neuroretinal fluorescein angiography in patients with Fabry disease and compare these to renal (measured by GFR).

Specific Aim 3. To show that the change in capillary perfusion studies when compared to baseline in response to enzyme replacement therapy treatment over time, as a manifestation of tissue burden and prognosis is a more sensitive biomarker of the extent of patient disease than corneal keratopathy.

ELIGIBILITY:
Inclusion Criteria:

* Fabry patient
* evidence of angiopathy (renal, cardiac, or ocular)
* Patients above the age of 18

Exclusion Criteria:

* Patients unable or unwilling to provide written informed consent will not be recruited
* Patients who are below the age of 18
* Patients who have not or will not be undergoing Fluorescein angiography
* Allergy to fluorescein
* Pregnant women and fetuses are exclude from the study due to risks related to fluorescein and no direct benefit to the pregnant woman and fetus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Initially any Fabry patient, age 18 and above who has a confirmed diagnosis of Fabry disease by previously identifying plasma or leukocyte α-galactosidase A (α-gal A) deficiency, will be recruited from all participating physician practices. Those who present with evidence of angiopathy (with specific attention to the target organs: renal, cardiac, or ocular) will be recruited for the study.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2010-07; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Presence of specific findings commonly associated with Fabry's disease using neuroretinal examination | every 6 months, for up to 3 years

SECONDARY OUTCOMES:
Capillary perfusion abnormalities in optic nerve and retina | every 6 months, for up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Deborah M Grzybowski, PhD, Principal Investigator — Ohio State University
Locations (1):
- Eye and Ear Institute, Columbus, Ohio, United States

REFERENCES:
- [Background] Caggana M, Ashley GA, Desnick RJ, Eng CM. Fabry disease: molecular carrier detection and prenatal diagnosis by analysis of closely linked polymorphisms at Xq22.1. Am J Med Genet. 1997 Aug 22;71(3):329-35. PMID 9268104
- [Background] Eng CM, Fletcher J, Wilcox WR, Waldek S, Scott CR, Sillence DO, Breunig F, Charrow J, Germain DP, Nicholls K, Banikazemi M. Fabry disease: baseline medical characteristics of a cohort of 1765 males and females in the Fabry Registry. J Inherit Metab Dis. 2007 Apr;30(2):184-92. doi: 10.1007/s10545-007-0521-2. Epub 2007 Mar 8. PMID 17347915
- [Background] Wilcox WR, Oliveira JP, Hopkin RJ, Ortiz A, Banikazemi M, Feldt-Rasmussen U, Sims K, Waldek S, Pastores GM, Lee P, Eng CM, Marodi L, Stanford KE, Breunig F, Wanner C, Warnock DG, Lemay RM, Germain DP; Fabry Registry. Females with Fabry disease frequently have major organ involvement: lessons from the Fabry Registry. Mol Genet Metab. 2008 Feb;93(2):112-28. doi: 10.1016/j.ymgme.2007.09.013. Epub 2007 Nov 26. PMID 18037317
- [Background] Glass RB, Astrin KH, Norton KI, Parsons R, Eng CM, Banikazemi M, Desnick RJ. Fabry disease: renal sonographic and magnetic resonance imaging findings in affected males and carrier females with the classic and cardiac variant phenotypes. J Comput Assist Tomogr. 2004 Mar-Apr;28(2):158-68. doi: 10.1097/00004728-200403000-00002. PMID 15091117
- [Background] Eng CM, Germain DP, Banikazemi M, Warnock DG, Wanner C, Hopkin RJ, Bultas J, Lee P, Sims K, Brodie SE, Pastores GM, Strotmann JM, Wilcox WR. Fabry disease: guidelines for the evaluation and management of multi-organ system involvement. Genet Med. 2006 Sep;8(9):539-48. doi: 10.1097/01.gim.0000237866.70357.c6. PMID 16980809
- [Background] Svarstad E, Bostad L, Kaarboe O, Houge G, Tondel C, Lyngdal PT, Iversen BM. Focal and segmental glomerular sclerosis (FSGS) in a man and a woman with Fabry's disease. Clin Nephrol. 2005 May;63(5):394-401. doi: 10.5414/cnp63394. PMID 15909601
- [Background] Tondel C, Bostad L, Hirth A, Svarstad E. Renal biopsy findings in children and adolescents with Fabry disease and minimal albuminuria. Am J Kidney Dis. 2008 May;51(5):767-76. doi: 10.1053/j.ajkd.2007.12.032. Epub 2008 Mar 20. PMID 18436087
- [Background] Tondel C, Bostad L, Laegreid LM, Houge G, Svarstad E. Prominence of glomerular and vascular changes in renal biopsies in children and adolescents with Fabry disease and microalbuminuria. Clin Ther. 2008;30 Suppl B:S42. doi: 10.1016/s0149-2918(08)80036-7. No abstract available. PMID 18395135
- [Background] Tondel C, Laegreid LM, Hirth A, Houge G, Mansson JE, Sovik O. [Intravenous enzyme substitution therapy in children with Fabry's disease]. Tidsskr Nor Laegeforen. 2003 Dec 4;123(23):3388-90. Norwegian. PMID 14713976
- [Background] Strujic BJ, Jeren T. Fabry disease--a diagnostic and therapeutic problem. Ren Fail. 2005;27(6):783-6. doi: 10.1080/08860220500244856. PMID 16350834
- [Background] Gilbert-Barness E. Review: Metabolic cardiomyopathy and conduction system defects in children. Ann Clin Lab Sci. 2004 Winter;34(1):15-34. PMID 15038665
- [Background] Kampmann C, Wiethoff CM, Perrot A, Beck M, Dietz R, Osterziel KJ. The heart in Anderson Fabry disease. Z Kardiol. 2002 Oct;91(10):786-95. doi: 10.1007/s00392-002-0848-5. PMID 12395219
- [Background] Whybra C, Kampmann C, Willers I, Davies J, Winchester B, Kriegsmann J, Bruhl K, Gal A, Bunge S, Beck M. Anderson-Fabry disease: clinical manifestations of disease in female heterozygotes. J Inherit Metab Dis. 2001 Dec;24(7):715-24. doi: 10.1023/a:1012993305223. PMID 11804208
- [Background] Mitsias P, Levine SR. Cerebrovascular complications of Fabry's disease. Ann Neurol. 1996 Jul;40(1):8-17. doi: 10.1002/ana.410400105. PMID 8687196
- [Background] Mehta A, Ginsberg L; FOS Investigators. Natural history of the cerebrovascular complications of Fabry disease. Acta Paediatr Suppl. 2005 Mar;94(447):24-7; discussion 9-10. doi: 10.1111/j.1651-2227.2005.tb02106.x. PMID 15895708
- [Background] Michels H, Mengel E. Lysosomal storage diseases as differential diagnoses to rheumatic disorders. Curr Opin Rheumatol. 2008 Jan;20(1):76-81. doi: 10.1097/BOR.0b013e3282f169fe. PMID 18281861
- [Background] Knowles SR, Weber EA, Berbrayer CS. Allergic reaction to fluorescein dye: successful one-day desensitization. Can J Ophthalmol. 2007 Apr;42(2):329-30. PMID 17392867
- [Background] Cook SC, Ferketich AK, Raman SV. Myocardial ischemia in asymptomatic adults with repaired aortic coarctation. Int J Cardiol. 2009 Mar 20;133(1):95-101. doi: 10.1016/j.ijcard.2007.12.015. Epub 2008 Feb 11. PMID 18262666